CLINICAL TRIAL: NCT03069742
Title: Web-based Decision Aids for Breast Cancer Risk Assessment and Increasing Breast Cancer Chemoprevention in the Primary Care Setting: Randomized Controlled Trial
Brief Title: Study of Web-based Decision Aids for Increasing Breast Cancer Chemoprevention in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine D. Crew, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAP4151 II; R01CA177995 (NIH)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer Prevention; Risk Assessment; Chemoprevention; Decision Making
MeSH Terms: conditions — Breast Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Experimental): Women at high risk for developing breast cancer will use a decision support tool, RealRisks, that facilitates discussion of breast cancer risk with their providers who will have access to the BNAV provider clinical decision support tool.
  Interventions: Other: RealRisks; Other: BNAV
- Control Group (No Intervention): Women at high risk for developing breast cancer will receive standard breast health education brochures.

INTERVENTIONS:
Other: RealRisks — RealRisks is a web-based patient decision aid with modules that present information about risk assessment and chemoprevention.
  Other Names: RealRisks patient-centered decision aid (DA)
  Arms: Decision Aid
Other: BNAV — Breast Cancer Risk Navigation (BNAV) tool is a web-based decision support tool with modules that present pertinent information for primary care providers regarding breast cancer risk assessment and preventative measures for their patients.
  Other Names: Breast Cancer Risk Navigation (BNAV) tool; BNAV provider clinical decision support tool
  Arms: Decision Aid

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to evaluate a decision support website (RealRisks) designed to inform patients about breast cancer prevention options. It is coupled with a physician-centered (BNAV) decision support website as part of clinical workflow in the primary care setting. The investigators hypothesize that improving accuracy of breast cancer risk perception and understanding of the risks and benefits of breast cancer risk lowering drugs, also known as chemoprevention, will increase the uptake of chemoprevention in the primary care setting.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women in the U.S. and the primary prevention of this disease is a major public health issue. The U.S. Preventive Services Task Force and other professional organizations recommend that clinicians discuss chemoprevention with high-risk women. Breast cancer chemoprevention with anti-estrogens, such as tamoxifen, raloxifene, exemestane, and anastrozole, is under-utilized, despite several randomized controlled trials demonstrating a 40-65% decrease in breast cancer incidence among high-risk women. Compounding this underutilization is the fact that a large proportion of women may be unaware of their high-risk status due to the investigators' inability to adequately screen them in the primary care setting. Further research is needed to determine how knowledge about breast cancer, actual/perceived risk, and risks/benefits of chemoprevention are best communicated to women in order to promote breast cancer prevention strategies.

The investigators hypothesize that combining a patient-centered decision aid with a physician-centered decision support tool integrated into clinic workflow will improve accuracy of breast cancer risk perception, facilitate referrals for specialized risk counseling, and increase chemoprevention uptake. We anticipate that the BNAV tool will facilitate referrals to the breast clinic by primary care providers (PCPs) and that the RealRisks decision aid will prime high-risk women to seek these referrals. The primary endpoint is uptake of a selective estrogen receptor modulator (SERM) or Aromatase inhibitor (AI) for breast cancer chemoprevention at 6 months (after the next primary care appointment) in the active arm compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* 5-year breast cancer risk ≥ to 1.67% or lifetime risk ≥ to 20% according to the Gail risk model; or a 5-year breast cancer risk ≥ 1.67% according to the Breast Cancer Surveillance Consortium (BCSC) model
* The participant understands and is willing to provide informed consent in English or Spanish
* Has a primary care provider at Columbia University Medical Center (CUMC) / New York-Presbyterian Hospital

Exclusion Criteria:

* Prior use of a selective estrogen receptor modulator (SERM) or aromatase inhibitor (AI) for chemoprevention
* Prior history of breast cancer

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Chemoprevention uptake rate among high-risk women | 6 months (after the next primary care visit)
  The primary endpoint is to determine the uptake rate of a SERM or AI medication for breast cancer chemoprevention at 6 months (after the next primary care visit) in the active arm compared to usual care (control arm). Electronic health records will be used to track chemoprevention uptake after exposure to the intervention, the RealRisks decision aid, or the control, standard standard breast health education brochures.

SECONDARY OUTCOMES:
Chemoprevention intention rate among high-risk women (Likert Scale Score) | 1 month
  Behavioral intention for chemoprevention will be assessed one month after baseline among those in the active arm compared to patients receiving usual care (control arm).
High-risk referral rates to the breast clinic | 6 months (after the next primary care visit)
  To study appropriate referral rate to the breast clinic by primary care providers of high-risk patients in the active arm compared to patients receiving usual care (control arm).
Completion of high-risk consultations at the breast clinic | 6 months (after the next primary care visit)
  To study appointment completion rate at the breast clinic by high-risk patients in the active arm compared to patients receiving usual care (control arm).

OTHER OUTCOMES:
Change in the accuracy of risk perception (Likert Scale Score) | 6 months
  To measure the patient's accuracy of perceived breast cancer risk before and after exposure to the RealRisks decision aid compared to those patients in the control group receiving usual care. Perception will be assessed by comparing the difference between a patient's perceived risk and their actual risk based on the Gail breast cancer model. Patients are asked to make a comparative risk assessment about themselves on a 3-point Likert scale.
Change in a patient's breast cancer knowledge (Survey Score) | 6 months
  To assess patient's breast cancer knowledge before and after exposure to the RealRisks decision aid compared to those patients in the control arm by comparing the difference between a patient's responses to a 13-item scale assessing knowledge with response options of true, false, or unsure.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Crew, MD, MS, Principal Investigator — Columbia University; Rita Kukafka, DrPH, MA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kukafka R, Yi H, Xiao T, Thomas P, Aguirre A, Smalletz C, David R, Crew K. Why Breast Cancer Risk by the Numbers Is Not Enough: Evaluation of a Decision Aid in Multi-Ethnic, Low-Numerate Women. J Med Internet Res. 2015 Jul 14;17(7):e165. doi: 10.2196/jmir.4028. PMID 26175193
- [Background] Yi H, Xiao T, Thomas PS, Aguirre AN, Smalletz C, Dimond J, Finkelstein J, Infante K, Trivedi M, David R, Vargas J, Crew KD, Kukafka R. Barriers and Facilitators to Patient-Provider Communication When Discussing Breast Cancer Risk to Aid in the Development of Decision Support Tools. AMIA Annu Symp Proc. 2015 Nov 5;2015:1352-60. eCollection 2015. PMID 26958276
- [Derived] Crew KD, Silverman TB, Vanegas A, Trivedi MS, Dimond J, Mata J, Sin M, Jones T, Terry MB, Tsai WY, Kukafka R. Study protocol: Randomized controlled trial of web-based decision support tools for high-risk women and healthcare providers to increase breast cancer chemoprevention. Contemp Clin Trials Commun. 2019 Aug 22;16:100433. doi: 10.1016/j.conctc.2019.100433. eCollection 2019 Dec. PMID 31497674
- See also: Pre-screening questionnaire — http://bit.ly/BCpreventionstudy